CLINICAL TRIAL: NCT07047716
Title: A Phase 3, Single-Arm Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Once-Yearly Intramuscular Lenacapavir for HIV Pre-exposure Prophylaxis (PrEP) in People With an Indication for PrEP
Brief Title: Study of Lenacapavir as a Once-Yearly Injection for HIV Pre-exposure Prophylaxis (PrEP)
Acronym: PURPOSE 365
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GS-US-712-7286
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV Pre-exposure Prophylaxis
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Intervention Model Description: It is a single arm study that means all participants will receive LEN. However, the study provides LEN in 2 phases, therefore, the two phases are reported as 2 separate arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenacapavir (LEN) (Experimental): Participants with an indication for pre-exposure prophylaxis will receive for approximately 52 weeks:
  * LEN 3000 mg injection once on Day 1
  * Oral LEN 600 mg on Day 1 and Day 2 during the Main Study Period
  Participant will receive additional oral LEN if IM injection are not available.
  Interventions: Drug: Lenacapavir Injection; Drug: Lenacapavir Tablet
- LEN Extension Phase (Experimental): Participants with an indication for pre-exposure prophylaxis will receive LEN 3000 mg injection once on Day 1 (approximately one year after their initial dose) during the Extension Phase.
  Participants will receive oral LEN if IM injections are not available.
  Interventions: Drug: Lenacapavir Injection; Drug: Lenacapavir Tablet

INTERVENTIONS:
Drug: Lenacapavir Injection — Administered intramuscularly
Drug: Lenacapavir Tablet — Administered orally

SUMMARY:
The goal of this clinical study is to learn more about the study drug lenacapavir (LEN), safety, tolerability, and pharmacokinetics (how LEN is absorbed, modified, distributed, and removed from the body of the participants) of once-yearly intramuscular for HIV pre-exposure prophylaxis (PrEP) in people with an indication for PrEP.

The primary objective of this study is to evaluate the pharmacokinetics (PK) and the safety and tolerability of intramuscular (IM) every 12 months (Q12M) LEN for PrEP among people with an indication for PrEP.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 16 years of age at screening.
* Receptive anal or vaginal sex in the past 6 months and at least 1 of the following:

  1. Condomless receptive sex (vaginal or anal) with 1 or more sex partners of unknown HIV status during the past 6 months
  2. For a person who has engaged in anal sex in the past 6 months: diagnosis of syphilis, gonorrhea, or chlamydia in the past 6 months
  3. For a person who has engaged in vaginal sex in the past 6 months: diagnosis of syphilis or gonorrhea in the past 6 months
  4. Sex with partner known to be living with HIV with an unknown or detectable viral load in the past 6 months
* Negative local rapid fourth generation HIV-1/2 antibody (Ab)/antigen (Ag) test, central fourth generation HIV-1/2 Ab/Ag, and HIV-1 RNA quantitative nucleic acid amplification testing (NAAT) at screening.

Key Exclusion Criteria:

* Current signs or symptoms suggesting HIV infection
* Acute viral hepatitis A, B, or C or evidence of chronic hepatitis B or C infection
* Severe hepatic impairment or a history of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, variceal bleeding)
* Past or current participation in HIV vaccine or HIV broadly neutralizing antibody study unless participant provides documentation of receipt of placebo (ie, not active product)
* Prior use of oral LEN in the past 90 days or subcutaneous LEN in the past 18 months

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender men, Transgender women, Transgender men, Cisgender women, and Gender non-binary
Enrollment: 300 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Plasma LEN Ctrough at Week 52 | Week 52
  Ctrough is defined as the concentration at the end of the dosing interval.
Percentage of Participants Experiencing Treatment-emergent Adverse Event (TEAEs) | First dose up to 30 days post last dose (approximately 3 years)
Percentage of Participants Experiencing Treatment-emergent Clinical Laboratory Abnormalities | First dose up to 30 days post last dose (up approximately 3 years)
Percentage of Participants With Discontinuation due to Adverse Event | First dose up to 30 days post last dose (approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (31):
- United States (31):
  - UAB Sexual Health Research Clinic, Birmingham, Alabama
  - UCLA Clinic Care, Los Angeles, California
  - Ruane Clinical Research Group, Inc., Los Angeles, California
  - UCLA Vine Street Clinic, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - BIOS Clinical Research, Palm Springs, California
  - UCSD AntiViral Research Center (AVRC), San Diego, California
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - Yale University; School of Medicine; AIDS Program, New Haven, Connecticut
  - Whitman-Walker Institute, Inc., Washington D.C., District of Columbia
  - Children's National Hospital, Washington D.C., District of Columbia
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - The ID Prevention Research Unit, Miami, Florida
  - University of South Florida - Curran Children's Health Center, Tampa, Florida
  - The Hope Clinic of Emory University, Atlanta, Georgia
  - Ponce de Leon Center Clinical Research Site, Atlanta, Georgia
  - University of Illinois-Chicago (UIC), Center for Dissemination and Implementation Sciences (CDIS), Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - University Medical Center, New Orleans, Louisiana
  - Johns Hopkins Hospital - Clinical Research Unit, Baltimore, Maryland
  - Fenway Health, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Icahn School of Medicine at Mount Sinai - Clinical and Translational Research Center, New York, New York
  - ICAP at Columbia University- Bronx Prevention Center, The Bronx, New York
  - NC TraCS Institute - CTRC, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Penn Prevention Unit, Philadelphia, Pennsylvania
  - Philadelphia FIGHT Community Health Centers, Jonathan Lax Treatment Center, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - The Crofoot Research Center, Houston, Texas
  - Vaccine Trials Unit - Fred Hutchinson Cancer Center / University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07047716